CLINICAL TRIAL: NCT06090942
Title: The Effectiveness of Cognitive Training for Digital Biomarkers: Evidence From the Urban and Rural Area
Brief Title: Cognitive Training for Digital Biomarkers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Huie-Ling Chiu, Associate professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: N202303103
Record Dates: First submitted 2023-08-16; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Cognitive Decline; Healthy Aging
Keywords: digital biomarker
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive training (Experimental): Smartphone-based cognitive training
  Interventions: Other: Smartphone-based cognitive training
- Usual care (No Intervention): No intervention

INTERVENTIONS:
Other: Smartphone-based cognitive training — Smartphone-based cognitive training
  Arms: Cognitive training

SUMMARY:
This study aims to conduct cognitive training for digital biomarkers among older adults.

DETAILED DESCRIPTION:
The prevalence of dementia in rural areas is higher than in urban areas. However, the resource and research input on cognitive training for rural older adults still needs improvement. There is also no solution for preventing or early detection of dementia in rural areas. Unlike biomarkers that require invasive detection, digital biomarkers have been advocated in recent years for early disease prediction. However, there are still few studies on the effectiveness of digital biomarkers in evaluating cognitive function in the elderly. In addition, although previous studies have confirmed that cognitive training can be effective for older adults, it is difficult for the elderly in rural areas to obtain these cognitive-promoting resources due to distance. Moreover, the autonomy and right of choice of older adults are the keys to the success of their health behavior change.

ELIGIBILITY:
Inclusion Criteria:

1. At least 60 years of age, Can communicate in Chinese (Taiwanese)
2. Bring your own mobile device with Internet access.
3. Can act alone without physical impairment；full score of basic activities of daily living scale and instrumental activities of daily living scale.

Exclusion Criteria:

1. Dementia diagnosed by a physician and in compliance with ICD-10
2. Physician diagnosed with significant mental illness or communication impairment
3. Participated in other cognitive training studies within the past year
4. Medical conditions associated with rapid functional and cognitive decline
5. Severe visual impairment

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
digital biomarker | pretest, immediate post test, 3 month follow-up, 6 month follow-up
  wearable device of stress and sleep, EEG power in alpha band, Delta and Theta frequency-bands

SECONDARY OUTCOMES:
Montreal Cognitive Assessment(MoCA) | pretest, immediate post test, 3 month follow-up, 6 month follow-up
  The Montreal Cognitive Assessment (MoCA) is a cognitive screening tool designed to identify mild cognitive impairment, providing a quick assessment of different cognitive domains including memory, attention, language, and executive functions. It is widely utilized in clinical and research settings.The MoCA is scored out of a maximum of 30 points. A score of 26 and above is generally considered to be normal, although the specific cutoff can depend on the individual's age, educational level, and other demographic factors.
Digit Span(DS) | pretest, immediate post test, 3 month follow-up, 6 month follow-up
  Digit Span (DS) is a common test used in neuropsychological assessments to measure working memory, attention, and concentration. Each correctly repeated sequence yields one point. There are typically 16 items for the Forward Digit Span. The Backward Digit Span also has 16 items.
Digit Vigilance Test(DVT) | pretest, immediate post test, 3 month follow-up, 6 month follow-up
  The Digit Vigilance Test (DVT) is a psychological assessment tool used to measure attention and concentration, mainly focused on visual scanning and processing speed. The number of correct identifications and the time taken to complete the task are typically measured.
Computerized version of Wisconsin Card Sort Test (WCST) | pretest, immediate post test, 3 month follow-up, 6 month follow-up
  The Wisconsin Card Sorting Test (WCST) is a well-established neuropsychological test widely used to assess executive functions, mainly focusing on abstract reasoning and the ability to shift cognitive strategies in response to changing environmental contingencies (i.e., set-shifting or cognitive flexibility). The computerized version of the WCST allows for efficient, standardized administration and scoring, often reducing examiner bias and error.
Stroop color-word test (SCWT) | pretest, immediate post test, 3 month follow-up, 6 month follow-up
  The Stroop Color-Word Test (SCWT) evaluates cognitive processing speed, selective attention, and cognitive flexibility, which are aspects of executive functioning. It's particularly notable for its ability to detect cognitive interference and inhibition control.Scores are typically based on:Correct Responses, Time Taken, Error Rate and Interference Score.

IPD SHARING:
Plan to Share IPD: No